CLINICAL TRIAL: NCT06071364
Title: Morphological Changes in Selected Back Muscles and Their Association With Back Extensors Strength in Subjects With Chronic Non-Specific Low Back Pain
Brief Title: Morphological Changes in Back Muscles With Low Back Pain Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: omnia Yasser Mohamed Talat Harb (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, omnia Yasser Mohamed Talat Harb, principal investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/004639
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Chronic Non-specific Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic nonspecific low back pain patients: Twenty-nine participants experienced chronic non-specific low back pain for over three months without any referred pain in their legs.
  Interventions: Diagnostic Test: Ultrasonography imaging and Hand-held dynamometer (HHD)
- Asymptomatic subjects: Twenty-nine subjects without symptoms of low back pain
  Interventions: Diagnostic Test: Ultrasonography imaging and Hand-held dynamometer (HHD)

INTERVENTIONS:
Diagnostic Test: Ultrasonography imaging and Hand-held dynamometer (HHD) — Ultrasound imaging system will be used to evaluate the thickness, cross -sectional area and fat infiltration of lumbar extensors lumbar multifidus , erector spinae and quadratus lumborum muscles.
  The hand-held dynamometer assessing isometric lumbar muscles strength

SUMMARY:
The purpose of this study is to assess the morphological changes in the lumbar multifidus, Erector spinae and Quadratus lumborum muscles and to investigate whether they are correlated with trunk extensor muscle strength in CNSLBP subjects.

and to compare between these morphological changes during rest and contraction and to compare these results with control group.

Twenty-nine subjects with CNSLBP and 29 age-matched healthy controls will be assessed by ultrasonography to detect the morphological changes of these muscles during rest and contraction ,and assessed strength of back extensors by hand-held dynamometer, and assessed functional disability by Arabic version of Oswestry disability index . They will be asked to sign the informed consent form.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common musculoskeletal disorders leading to inactivity, postural disorders, and muscle problems and can result in disability, reduced quality of life, and workforce loss.

Low back pain is commonly classified as non-specific (90%) or specific (10%) according to reported cause and as acute (<6 weeks), subacute (6-12 weeks) or chronic (more than12 weeks) according to duration of symptoms.

Many factors have been reported to play a role in the etiology of Chronic non-specific Low back pain (CNSLBP) including occupational factors, personal factors, and behavioral risk factors. In addition, recent studies associate low back pain with physical factors such as lumbar spinal stiffness, muscle shortness, and decreased endurance and muscle strength.

Many studies have mainly focused on the morphological aspects of paraspinal muscles including lumbar multifidus , Erector spinae and Quadratus lumborum muscles, which play an essential role in patients with CNSLBP in terms of functional disability and the planning of rehabilitation modalities.

Twenty-nine subjects with CNSLBP and 29 age-matched healthy controls will be recruited through direct referral. They will be asked to sign the informed consent form.

To authors knowledge no previous research had investigated the correlation between morphological changes and strength of back muscles in subjects with CNSLBP

The finding of this proposed work may help researchers interested in CNSLBP's etiology and natural course which can be considered a topic that are still poorly understood. To reduce the occurrence and severity of CNSLBP, it is essential to help understand its cause and determine whether there are any risk factors that may be changed.

The finding of this proposed work may benefit patients diagnosed with CNSLBP. If the diagnosis of back pain, function, and muscle strength in those patients become more clear , not only this may make them return to work early but may also improve psychological status.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both genders with CNSLBP (pain> 3 months)
2. The subject's age ranged between 18 and 45.
3. waist-to-height ratio (WHtR) < 0.5 or = 0.5

Exclusion Criteria:

1. Untreated neurological and/or mental illness
2. History of trauma in the last 6 months.
3. Sacroiliac joint pathologies.
4. Spinal fracture or dislocation.
5. Spinal instability (e.g., spondylolisthesis or retrolisthesis)
6. Sensitivity to ultrasound gel diagnosed by a medical doctor.
7. Serious musculoskeletal problems or other pathologies.
8. Previous surgery in lower limb(s)
9. Females during Pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Outpatient clinic of Mallawi Hospital
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Functional disability | from 5 to 10 minutes
  Functional disability will be measured by Arabic version of Oswestry Disability Index (ODI). The ODI is a 10-item self-assessing questionnaire, each item contains 6 levels of answers that can be scored from 0 (minimum degree of difficulty in that activity) to 5 (maximum degree of difficulty). These items are pain, personal care, lifting and moving objects, walking, sitting, standing, sleep disorders caused by the low back pain, sex life, social life, and traveling The Arabic version of ODI has been established as a valid measure, and demonstrated excellent intra-observer reliability.
Back muscle strength | from 5 to 7 minutes
  will be measured by Hand-held dynamometer (HHD): assessing isometric lumbar muscles strength. In a clinical setting, it is viewed as easy to use, portable and cost-effective for the precise measurement of lumbar muscles strength. Intra-rater and inter-rater reliability of hand-held dynamometer for assessing isometric lumbar muscle strength in asymptomatic healthy population showed an excellent intra-rater (ICC 2, k = 0.95 to 0.97) and inter-rater (ICC 2, k = 0.94 to 0.95) .
Muscle Thickness | about 15 minutes
  evaluate the thickness of lumbar extensors lumbar multifidus, erector spinae and quadratus lumborum muscles and will be assessed by an experienced and qualified radiologist using US unit at rest and contraction on both right and left sides.
Muscle Cross Sectional Area | about 15 minutes
  evaluate cross -sectional area of lumbar extensors lumbar multifidus, erector spinae and quadratus lumborum muscles and will be assessed by an experienced and qualified radiologist using US unit during rest and contraction on both right and left sides.
Muscle Fat infiltration | about 15 minutes
  evaluate Fat infiltration of lumbar extensors lumbar multifidus, erector spinae and quadratus lumborum muscles and will be assessed by an experienced and qualified radiologist using US unit during rest and contraction on both right and left sides.

CONTACTS AND LOCATIONS:
Overall Officials: omnia yasser, master, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
undecided